CLINICAL TRIAL: NCT01578408
Title: Corail-SP Study - A Prospective Randomized Comparison Between Cemented and Uncemented Hydroxyapatite Coated Prosthesis Stems in Total Hip Arthroplasty in Patients With Femoral Neck Fractures
Brief Title: Cemented Versus Uncemented Stems in Total Hip Arthroplasty in Patients With Femoral Neck Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Arun Patel, MD, Senior Physician in Orthopaedic Surgery, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Corail-SP Study
Record Dates: First submitted 2012-04-11; First posted 2012-04-17 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral neck fractures; Uncemented; Hydroxyapatite; Coated; Femoral; Stems; Hip fractures; THA; THR; Cemented; Fat embolism; Cognition; Inflammatory response; Mobilization
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures; Embolism, Fat | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uncemented HA Coated Corail stem (Active Comparator): Surgery with an inversed hybrid arthroplasty with an uncemented hydroxyapatite coated Corail stem and a cemented Marathon cup (DePuy).
  Interventions: Procedure: Total Hip Arthroplasty; Device: Uncemented HA Coated Corail stem
- Cemented Lubinus SPII stem (control arm) (Active Comparator): Surgery with a totally cemented option with a Lubinus SPII stem and a IP cup (Link).
  Interventions: Procedure: Total Hip Arthroplasty; Device: Cemented Lubinus SPII stem (control arm)

INTERVENTIONS:
Procedure: Total Hip Arthroplasty
Device: Cemented Lubinus SPII stem (control arm) — Cemented Lubinus femoral stem. Cemented IP acetabular cup. (Link).
  Arms: Cemented Lubinus SPII stem (control arm)
Device: Uncemented HA Coated Corail stem — Uncemented hydroxyapatite coated Corail femoral stem. Cemented Marathon acetabular cup. (DePuy).
  Arms: Uncemented HA Coated Corail stem

SUMMARY:
The purpose of this prospective randomized study is to compare the quality of treatment between cemented versus uncemented hydroxyapatite coated femoral stems in Total Hip Arthroplasty (THA) in patients who suffers from dislocated femoral neck fractures.

Our hypothesis is that an uncemented option spares the patient the operative load of the cementing procedure, i e risk of fatty embolism and inflammatory response, which in turn also perhaps reduces the postoperative cognition strain and improves mobilization parameters.

If the uncemented option has the same excellent fixation in poor bone stock, as in the case of these osteopenic fractures, and also has the same good clinical outcome, it would be a viable standard option for the treatment of dislocated femoral neck fractures.

DETAILED DESCRIPTION:
Corail-SP study. A prospective randomized study to compare the quality of treatment between cemented versus uncemented hydroxyapatite coated femoral stems in Total Hip Arthroplasty (THA) in patients who suffers from dislocated femoral neck fractures.

Femoral neck fractures often occurs among the fragile elderly patients who have a higher degree of co-morbidity. The 3-month mortality is 13%. The incidence of risk of fracture complications when using osteosyntheses are as high as 30-40%, mainly due to non union, which leads to impairments in quality of life, locomotion and pain.

For that reason more patients nowadays are submitted to a cemented hemiarthroplasty or a total hip arthroplasty directly after their injury - at the same time the problem with fatty embolism syndrome has been recognized. When cementing during surgery, the bone marrow is pushed into the blood stream, which can affect the cardiopulmonary function and even the mental functions.

As a measure for reducing those risks an uncemented hip arthroplasty is sometimes used instead.

The pros and cons with uncemented fixation is poorly examined which this study will try to scrutinize.

100 patients with dislocated (Garden classification III-IV) femoral neck fractures who have the clinical indication of undergoing a Total Hip Arthroplasty are asked and included at Mölndals Hospital (part of Sahlgrenska University Hospital).

Randomization to either; an inversed hybrid arthroplasty with an uncemented hydroxyapatite coated Corail stem and a cemented Marathon cup (DePuy), alternatively to, a totally cemented option with a Lubinus SPII stem and a IP cup (Link).

Preoperatively:

Patient questionnaires regarding cognitive and social status, hip function, quality of life (QoL), activity level. Standard hip and pelvis X-ray. Blood sample for biomarkers.

Peroperatively:

Pulmonary artery catheter measurements of pulmonary artery pressure, cardiac output, ejection fraction of the right ventricle. Surgeon's questionnaire regarding prosthesis components, duration of surgery, blood group, bleeding volume, oxygen saturation. Half of the patients are marked with tantalum pellets for radiostereometric analysis (RSA). Biomarkers.

Postoperatively:

Standard X-ray. On the patients marked with tantalum pellets RSA is performed. Bone density scan (DXA). Measurements regarding cognition, ADL, mobilization. Eventual confusion is noted. Biomarkers every second day until discharge from hospital. Eventual wound infections or thromboembolic episodes are noted.

Follow up:

Outpatient return visits to physician 3, 6 months, 1, 2, 5, 7, 10 years postoperatively. Standard X-ray, RSA, DXA, Patient questionnaires regarding patient's satisfaction, QoL, activity level, hip function. Biomarkers.

Eventual gains with an uncemented prosthesis:

Reduced fatty embolism risk, reduced inflammatory response, reduced generalized symptoms/confusion, faster mobilization, shorter surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are acutely admitted to hospital with dislocated femoral neck fractures, that in clinical praxis are in the need of hip prosthesis surgery, are recruited in the study. The fracture shall not engage the lesser nor the greater trochanters.
* Patients who wants to participate in the study and who can consider participation for at least 1 year.
* Coming from independent dwelling conditions.
* Not dementia.
* Circa 60-85 years of age.
* Circa 50 patients in each arm/group shall be included at Mölndal's Hospital (part of Sahlgrenska University Hospital).

Exclusion Criteria:

* Patients who have difficulties in understanding the intent of the study.
* Rheumatic disorders (RA, Bechterew, SLE).
* Cortison treatment.
* Stroke with remaining weakness or neurological disorders with affection of locomotion.
* Dementia.
* Grave obesity with BMI >=30-35.
* Delay between time of injury and time of surgery exceeding 72 hours.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Time to mobilization. | During hospital stay, an expected average of 10 days.
  Time (days) to mobilization defined as independent walking with or without walking aids measured by ward physiotherapist with Traffic Light System and Sahlgrenska University Hospital Hip Score (SUHS).

SECONDARY OUTCOMES:
Cognitive status. Eventual confusion. | During hospital stay, an expected average of 10 days.
  Cognitive status measured once daily with Pfeiffer's test (Short Portable Mental Status Questionnaire - SPMSQ).
  Eventual confusion is noted once daily.
Oxygen saturation levels peroperatively. | Peroperatively (during surgery), an expected average of 2 hours.
  POX-measurements during different phases of surgery along with pulmonary catheter readings.
Bone remodeling around the hip prosthesis. | Postoperatively in average after 2 days. All follow up visits at 3, 6 months, 1, 2, 5, 7, 10 years.
  Measurements with hip DXA.
Biomarkers / inflammatory response. | Preoperatively in average 4 hours. Peroperatively at end of wound closure. Postoperatively 1, 3, 5, 7 days. All follow up visits at 3, 6 months, 1, 2, 5, 7, 10 years.
  Blood samples for measurement of the inflammatory response with biochip multi-array technology.
Fixation / migration / loosening of the hip prosthesis components. | Postoperatively in average after 2 days. All follow up visits at 3, 6 months, 1, 2, 5, 7, 10 years.
  Measured by radiostereometric analysis (RSA) in addition to the conventional pelvis and hip X-ray exams. Early radiological loosening of one or both of the prosthesis components is identified at an early stage with RSA.
Reoperation. | Postoperatively up to 10 years.
  In case of for example infection or dislocation.
PROM - Patient Reported Outcome Measurements. | Preoperatively in average 4 hours. Postoperatively at discharge from hospital at an expected average of 10 days. All follow up visits at 3, 6 months, 1, 2, 5, 7, 10 years.
  Questionnaires regarding Patient's satisfaction, Quality of life (EQ-5D), Activity level (UCLA), Harris Hip Score.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Kärrholm, Prof MD PhD, Study Director — Orthopaedic Department, Sahlgrenska University Hospital, Gothenburg, SWEDEN
Locations (1):
- Mölndals Hospital (part of Sahlgrenska University Hospital), Mölndal, Sweden